CLINICAL TRIAL: NCT00077623
Title: A Randomized, Controlled, Open-Label, Multi- Center, Parallel-Group Study to Demonstrate the Efficacy and Safety of RO0503821 When Administered Subcutaneously for the Maintenance Treatment of Anemia in Patients With Chronic Kidney Disease Who Are on Dialysis
Brief Title: A Study of Subcutaneous Mircera for the Treatment of Anemia in Dialysis Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA16740
Record Dates: First submitted 2004-02-10; First posted 2004-02-13 (Estimated); Results first posted 2016-04-26 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-04

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa; continuous erythropoietin receptor activator

ARMS (3):
- RO0503821 (1x/2 Weeks) (Experimental): Eligible participants received RO0503821 (Mircera [methoxy polyethylene glycol-epoetin beta]) subcutaneously, once every two weeks for 52 weeks. Participants received a starting dose of RO0503821 60, 100, or 180 microgram (mcg) which was based on the epoetin dose of<8000, 8000-16000, or >16000 international units (IU)/week, administered during the week preceding the switch to the study drug.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta (Mircera)
- RO0503821 (1x/4 Weeks) (Experimental): Eligible participants received RO0503821 subcutaneously, once every four weeks for 52 weeks. Participants received a starting dose of RO0503821 120, 200, or 360 mcg which was based on the epoetin dose of<8000, 8000-16000, or >16000 IU/week administered during the week preceding the switch to the study drug.
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta (Mircera)
- Epoetin Reference (Active Comparator): Eligible participants received their ongoing weekly subcutaneous dose of epoetin alfa or beta one, two or three times weekly for 52 weeks .
  Interventions: Drug: epoetin alfa or beta

INTERVENTIONS:
Drug: epoetin alfa or beta — iv 3 times weekly, as prescribed
  Arms: Epoetin Reference
Drug: methoxy polyethylene glycol-epoetin beta (Mircera) — 60, 100 or 180 micrograms sc (starting dose) every 2 weeks
  Arms: RO0503821 (1x/2 Weeks)
Drug: methoxy polyethylene glycol-epoetin beta (Mircera) — 60, 100 or 180 micrograms sc (starting dose) every 4 weeks
  Arms: RO0503821 (1x/4 Weeks)

SUMMARY:
This study will assess the efficacy and safety of subcutaneous (sc) Mircera given as maintenance treatment for renal anemia in chronic kidney disease patients on dialysis who were previously receiving sc epoetin. The anticipated time on study treatment is 1-2 years and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* chronic renal anemia;
* on dialysis therapy for at least 12 weeks before screening;
* receiving sc epoetin for at least 8 weeks before screening.

Exclusion Criteria:

* women who are pregnant, breastfeeding or using unreliable birth control methods;
* administration of another investigational drug within 4 weeks before screening, or during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2004-03; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (84):
- United States (17):
  - Hot Springs, Arkansas
  - Los Angeles, California
  - Riverside, California
  - Sacramento, California
  - San Jose, California
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Brooklyn Center, Minnesota
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Toledo, Ohio
  - Portland, Oregon
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Morgantown, West Virginia
- Belgium (4):
  - Brussels
  - Edegem
  - Ghent
  - Hasselt
- Brazil (2):
  - Curitiba
  - São Paulo
- Czechia (3):
  - Brno
  - Ostrava
  - Pilsen
- Odense, Denmark
- Finland (3):
  - HUS
  - Tampere
  - Turku
- France (12):
  - Bayonne
  - Boulogne
  - Cabestany
  - Caen
  - Limoges
  - Nîmes
  - Pantin
  - Poitiers
  - Saint-Germain-en-Laye
  - Saint-Priest-en-Jarez
  - Thionville
  - Tours
- Germany (3):
  - Bad Hersfeld
  - Berlin
  - Kaiserslautern
- Hungary (4):
  - Budapest
  - Debrecen
  - Miskolc
  - Pécs
- Italy (6):
  - Cremona
  - Lecco
  - Mestre
  - Modena
  - Prato
  - Venezia
- Mexico (2):
  - Cuernavaca
  - Mexico City
- New Zealand (2):
  - Christchurch
  - Wellington
- Panama City, Panama
- Poland (4):
  - Gdansk
  - Kielce
  - Krakow
  - Wroclaw
- Ponce, Puerto Rico
- Durban, South Africa
- Spain (6):
  - Alcorcón
  - Barcelona
  - Madrid
  - Palma de Mallorca
  - Pamplona
  - Santiago de Compostela
- Sweden (2):
  - Huddinge
  - Karlstad
- Taiwan (2):
  - Taichung
  - Taipei
- Thailand (2):
  - Bangkok
  - Phitsanulok
- United Kingdom (6):
  - Belfast
  - Cambridge
  - Dundee
  - Exeter
  - Leicester
  - London

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 817 participants were enrolled in this study conducted from 03 March 2004 to 23 September 2005 at 92 centers worldwide.
Pre-assignment Details: A total of 572 participants were randomized, of which 1 participant did not received the study drug.
Groups:
- RO0503821 (1x/2 Weeks): Eligible participants received RO0503821 (Mircera [methoxy polyethylene glycol-epoetin beta]) subcutaneously, once every two weeks for 52 weeks. Participants received a starting dose of RO0503821 60, 100, or 180 microgram (mcg) which was based on the epoetin dose of<8000, 8000-16000, or >16000 international units per week (IU/week), administered during the week preceding the switch to the study drug.
- Epoetin Reference: Eligible participants received their ongoing weekly subcutaneous dose of epoetin alfa or beta one, two or three times weekly for 52 weeks.
Period: Overall Study
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin Reference
Started | 190 | 191 | 191
Completed | 154 | 148 | 159
Not Completed | 36 | 43 | 32
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 10 | 1
Not completed — Other-Non safety reason | 18 | 15 | 19
Not completed — Insufficient therapeutic response | 2 | 0 | 0
Not completed — Death | 12 | 18 | 11
Not completed — Failure to return | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis was done on safety population which included all participants who received at least one dose of study drug.
Groups:
- RO0503821 (1x/2 Weeks): Eligible participants received RO0503821 subcutaneously, once every two weeks for 52 weeks. Participants received a starting dose of RO0503821 60, 100, or 180 mcg which was based on the Epoetin dose of<8000, 8000-16000,or >16000 International units [IU]/Week, administered during the week preceding the switch to the study drug.
- Total: Total of all reporting groups
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin Reference | Total
Number analyzed (Participants) | 190 | 190 | 191 | 571
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (15.40) | 62.5 (15.16) | 60.4 (14.70) | 61.1 (15.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 73 | 81 | 236
  Male | 108 | 117 | 110 | 335

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin Concentration From Baseline to Evaluation Periods
Description: A time adjusted mean change in hemoglobin (Hb) concentration was calculated using an area under the curve (AUC) approach, for both periods separately. Change in Hb concentration between the baseline and evaluation periods was calculated by subtracting the calculated average baseline Hb value from the average evaluation period Hb value. All blood samples for Hb measurements were taken prior to study drug administration. Analysis used last observation carried forward (LOCF) for missing Hb values to correct for the impact of early dropouts. The baseline period is defined as Week -4 to Week -1. The evaluation period is defined as Week 29 to Week 36.
Time Frame: Baseline (Week -4 to Week -1) and Evaluation period (Week 29 to Week 36)
Population: The Per Protocol population included all randomized participants except those not meeting inclusion criterion related to stable baseline Hb values, inadequate iron status, hemoglobinopathies/hemolysis, RBC transfusion/blood loss, with <5 recorded Hb values during the evaluation period, with missing administrations of the study drug/ reference drug
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- RO0503821 (1x/2 Weeks): Eligible participants received RO0503821 subcutaneously, once every two weeks for 52 weeks. Participants received a starting dose of RO0503821 60, 100, or 180 mcg which was based on the epoetin dose of<8000, 8000-16000, or >16000 IU/week, administered during the week preceding the switch to the study drug.
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin Reference
Number analyzed (Participants) | 154 | 153 | 167
g/dL | -0.00 (0.96) | -0.11 (0.97) | -0.12 (1.04)
Statistical Analysis 1: Comparison: RO0503821 (1x/2 Weeks) vs Epoetin Reference; The non-inferiority test for treatment differences in Hb change from baseline, based on ANCOVA analysis with a non-inferiority limit of -0.75 g/dL (Per Protocol Population); Test type: Non-Inferiority or Equivalence — The two RO0503821 dosing schedules were compared separately to epoetin reference using ANCOVA, with Hb at BL and region as the covariates. The test for non-inferiority were based on the lower limit of the two-sided 97.5% confidence interval for the difference between the two groups. When the lower limit was greater than or equal to -0.75 g/dL, the RO0503821 groups were regarded as non-inferior to the epoetin reference group. The confidence level of 97.5% was chosen to adjust for multiplicity; p < 0.0001, ANCOVA, CI for difference between groups — The p-value for the non-inferiority test can be derived via the t-test; Mean Difference between groups = 0.141, 97.5% CI 2-sided [-0.098 to 0.380]
Statistical Analysis 2: Comparison: RO0503821 (1x/4 Weeks) vs Epoetin Reference; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The two RO0503821 dosing schedules were compared separately to epoetin reference using ANCOVA, with Hb at BL and region as the covariates. The test for non-inferiority were based on the lower limit of the two-sided 97.5% confidence interval for the difference between the two groups. When the lower limit was greater than or equal to -0.75 g/dL, the RO0503821 groups were regarded as non-inferior to the epoetin reference group. The confidence level of 97.5% was chosen to adjust for multiplicity; p < 0.0001, ANCOVA, CI for difference between groups — The p-value for the non-inferiority test can be derived via the t-test; Mean Difference between groups = -0.022, 97.5% CI 2-sided [-0.262 to 0.217]

2. Secondary Outcome: Number of Participants Maintaining Average Hb Concentration During the Evaluation Period Within +-1 g/dL of Their Average Baseline Hb Concentration
Description: All mean Hb values recorded during the evaluation period were calculated and subtracted from the mean baseline Hb value for each participant. The number of participants maintaining their average Hb within +/- 1 g/dL of their average baseline hemoglobin concentration is given. The evaluation period is defined as Week 29 to Week 36.
Time Frame: Evaluation period (Week 29 to Week 36)
Population: The Intent-to-Treat (ITT) population included all randomized participants.
Measure: Number; unit: participants
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin Reference
Number analyzed (Participants) | 164 | 168 | 176
participants | 124 | 111 | 127

3. Secondary Outcome: Number of Participants With Red Blood Cell Transfusions
Description: The number of participants who received RBC transfusions were reported.
Time Frame: Up to Week 36
Population: Safety population included all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin Reference
Number analyzed (Participants) | 190 | 190 | 191
participants | 12 | 20 | 19

4. Secondary Outcome: Number of Participants With Any Adverse Events, Any Serious Adverse Events, and Deaths
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to week 52
Population: Safety population included all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin Reference
Number analyzed (Participants) | 190 | 190 | 191
participants
  Any AE's | 171 | 177 | 167
  Any SAE's | 70 | 73 | 85
  Deaths | 13 | 18 | 12

5. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: A marked abnormality range was defined as above and/or below a value which was considered to be potentially clinically relevant. Marked laboratory abnormalities were analyzed according to the Roche specified limits for the reference range of the following laboratory parameters: White blood cells (WBC) (3.0- 18.0 10^9/L), platelets (100 - 550 10^9/L), alanine aminotransferase (ALAT) (0 - 110 units per liter [U/L]), alkaline phosphatase (ALP [0 - 220 U/L]), aspartate aminotransferase (ASAT) (0 - 80 U/L), albumin >= 30 g/L, phosphate (0.75 - 1.60 millimoles per liter [mmol/L]), potassium (2.9 - 5.8 mmol/L), glucose (2.80 - 11.10 mmol/L).
Time Frame: Up to week 52
Population: Safety population included all participants who received at least one dose of study drug. Maximum number of participants available at the time of assessment were denoted as 'n'.
Measure: Number; unit: participants
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin Reference
Number analyzed (Participants) | 189 | 189 | 188
participants
  Platelets, high; n=189,189, 188 | 0 | 1 | 1
  Platelets, low; n=189,189, 188 | 8 | 11 | 1
  RBC, high; n = 118, 112, 115 | 0 | 2 | 1
  RBC, low; n = 118, 112, 115 | 48 | 48 | 73
  WBC, high; n=189,189, 188 | 1 | 2 | 5
  WBC, low; n=189,189, 188 | 3 | 4 | 4
  ALAT, high; n=189,189, 188 | 6 | 11 | 6
  ALP, high; n=189,189, 188 | 5 | 8 | 11
  ASAT, high; n=185,189, 186 | 4 | 5 | 2
  Albumin, low; n=182,186, 185 | 16 | 20 | 17
  Phosphate, high; n=189,189, 188 | 84 | 78 | 82
  Phosphate, low; n=189,189, 188 | 14 | 17 | 18
  Potassium, high; n=189,189, 188 | 32 | 38 | 38
  Potassium, low; n=189,189, 188 | 1 | 4 | 1
  Glucose fasting, high; n=126,137, 124 | 1 | 2 | 2
  Glucose fasting, low; n=126,137, 124 | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure - at Weeks 36 and 52 in Hemodialysis Participants
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) was measured in sitting position before and after dialysis session in haemodialysis participants.
Time Frame: From Baseline (Week -4 to Week -1) to Week 36 and Week 52
Population: Safety population included all participants who received at least one dose of study drug. Maximum number of participants available at the time of assessment was denoted as 'n'.
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin Reference
Number analyzed (Participants) | 150 | 153 | 158
mmHG
  DBP- before dialysis (Week 36, n=150,153, 157) | 0 (12.2) | 0 (15.5) | 1 (14.6)
  DBP- before dialysis (Week 52, n= 143, 136, 144) | -1 (13.8) | -1 (11.1) | 2 (14.3)
  DBP - After dialysis (Week 36, n=150, 150, 157) | 1 (13.2) | -0 (17.3) | -1 (15.7)
  DBP - After dialysis (Week 52, n= 141, 136, 142) | 0 (15) | 0 (14.9) | 2 (15.6)
  SBP - before dialysis(Week 36, n=150, 153, 158) | 1 (22.1) | 4 (26.1) | -1 (22.7)
  SBP - before dialysis(Week 52, n=143, 136,144) | -1 (25.2) | 3 (23.1) | 1 (23.4)
  SBP - After dialysis (Week 36, n=150, 152, 158) | -1 (24.4) | -0 (27.1) | -2 (26.8)
  SBP - After dialysis (Week 52, n=141, 136, 142) | 1 (24.1) | -2 (23.4) | 2 (23.9)

7. Secondary Outcome: Change From Baseline in Pulse Rate at Weeks 36 and 52 in Hemodialysis Participants
Description: Pulse rate in beats per minute (BpM) was measured at each study visit, i.e., once a week during the dose titration and evaluation periods, once every two weeks during the long-term safety observation period and at the final visit. It was measured before blood sampling and RO0503821/epoetin administration and before the dialysis session in haemodialysis participants.
Time Frame: From Baseline (Week -4 to Week -1) to Week 36 and Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: BpM
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin Reference
Number analyzed (Participants) | 147 | 149 | 156
BpM
  Pulse rate (Week 36, n=147,149, 156 ) | -0 (11.8) | 1 (11.3) | -0 (12.0)
  Pulse rate (Week 52, n= 140, 135, 142) | -0 (10.6) | 1 (12.5) | -0 (12.3)

8. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure at Weeks 36 and 52 in Peritoneal Dialysis Participants
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) was measured in sitting position before and after dialysis session in peritoneal dialysis participants.
Time Frame: From Baseline (Week -4 to Week -1) to Week 36 and Week 52
Population: Safety population included all participants who received at least one dose of study medication. Maximum number of participants available at the time of assessment were analysed and reported.
Measure: Mean (Standard Deviation); unit: mm HG
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin Reference
Number analyzed (Participants) | 8 | 10 | 12
mm HG
  DBP (Week 36, n=7,10,12 ) | 2 (12.8) | -7 (13.9) | 2 (15.5)
  DBP (Week 52, n= 8, 9, 12) | 1 (10.3) | -8 (18.7) | 2 (18.5)
  SBP - (Week 36, n=7, 10, 12) | 3 (26.7) | -20 (33.5) | 7 (29)
  SBP - (Week 52, n=8, 9,12) | 4 (22.1) | -20 (36.9) | 12 (19.6)

9. Secondary Outcome: Change From Baseline in Pulse Rate - Peritoneal Dialysis Participants
Description: Pulse rate in BpM was measured at each study visit, i.e., once a week during the dose titration and evaluation periods, once every two weeks during the long-term safety observation period and at the final visit. It was measured before blood sampling and RO0503821/epoetin administration and before the dialysis session in peritoneal dialysis participants.
Time Frame: From Baseline (Week -4 to Week -1) to Week 36 and Week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: BpM
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin Reference
Number analyzed (Participants) | 147 | 149 | 156
BpM
  Pulse rate (Week 36, n=147,149, 156) | 1 (16.7) | 4 (12.2) | 6 (6.9)
  Pulse rate (Week 52, n= 140, 135, 142) | -3 (12.7) | 1 (7.8) | 2 (7.8)

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: Serious adverse events and non-serious adverse events are reported in safety analysis set, which consists of all participants who received at least one dose of study drug and had a safety assessment performed post baseline.
Arm/Group | RO0503821 (1x/2 Weeks) | RO0503821 (1x/4 Weeks) | Epoetin Reference
Serious Adverse Events (participants affected / at risk) | 70/190 | 73/190 | 85/191
Other Adverse Events (participants affected / at risk) | 113/190 | 131/190 | 111/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RO0503821 (1x/2 Weeks) (N=190) | RO0503821 (1x/4 Weeks) (N=190) | Epoetin Reference (N=191)
Pneumonia (Infections and infestations) | 5 | 5 | 8
Gangrene (Infections and infestations) | 2 | 1 | 2
Sepsis (Infections and infestations) | 2 | 3 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 0 | 1 | 4
Bronchitis Acute (Infections and infestations) | 1 | 2 | 1
Bronchopneumonia (Infections and infestations) | 0 | 4 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 1
Septic Shock (Infections and infestations) | 1 | 3 | 0
Catheter Related Infection (Infections and infestations) | 0 | 1 | 2
Peritonitis bacterial (Infections and infestations) | 2 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1 | 1
Infected skin ulcer (Infections and infestations) | 0 | 0 | 2
Urinary tract infection bacterial (Infections and infestations) | 0 | 2 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Arteriovenous fistula site infection (Infections and infestations) | 0 | 1 | 0
Arteriovenous graft site abscess (Infections and infestations) | 0 | 1 | 0
Arteriovenous graft site infection (Infections and infestations) | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1 | 0
Cellulitis gangrenous (Infections and infestations) | 0 | 1 | 0
Cellulitis of male external genital organ (Infections and infestations) | 0 | 0 | 1
Diabetic foot infection (Infections and infestations) | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1
Endocarditis (Immune system disorders) | 0 | 0 | 1
Escherichia infection (Infections and infestations) | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1
Hepatitis c (Infections and infestations) | 0 | 1 | 0
Herpes ophthalmic (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Intestinal gangrene (Infections and infestations) | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 1
Pneumonia chlamydial (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Scrotal abscess (Infections and infestations) | 1 | 0 | 0
Sepsis syndrome (Infections and infestations) | 1 | 0 | 0
Serratia sepsis (Infections and infestations) | 0 | 1 | 0
Staphylococcal abscess (Infections and infestations) | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 8 | 6
Cardiac arrest (Cardiac disorders) | 2 | 4 | 4
Cardiac failure congestive (Cardiac disorders) | 2 | 5 | 3
Angina pectoris (Cardiac disorders) | 2 | 3 | 2
Aortic valve stenosis (Cardiac disorders) | 1 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 2
Angina unstable (Cardiac disorders) | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 2
Bradyarrhythmia (Cardiac disorders) | 2 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 2
Coronary artery atherosclerosis (Cardiac disorders) | 0 | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 1
Pericarditis (Cardiac disorders) | 0 | 1 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1
Coronary artery dissection (Cardiac disorders) | 0 | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 1
Coronary artery thrombosis (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 4 | 3 | 3
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 4 | 0 | 0
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 2
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 1 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 1 | 0
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0
Bezoar (Gastrointestinal disorders) | 0 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Duodenitis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Erosive duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Peritoneal haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Atherosclerosis obliterans (Vascular disorders) | 2 | 1 | 1
Hypotension (Vascular disorders) | 0 | 4 | 0
Atherosclerosis (Vascular disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 1 | 0
Intermittent claudication (Vascular disorders) | 1 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 2
Peripheral occlusive disease (Vascular disorders) | 0 | 2 | 0
Circulatory collapse (Gastrointestinal disorders) | 0 | 1 | 0
Deep vein thrombosis (Gastrointestinal disorders) | 1 | 0 | 0
Diabetic vascular disorder (Vascular disorders) | 1 | 0 | 0
Iliac artery stenosis (Vascular disorders) | 0 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Peripheral embolism (Vascular disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 2 | 2
Toxic induced encephalopathy (Nervous system disorders) | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1
Brain stem haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Facial palsy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 1
Hypoxic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 1 | 0
Thrombotic stroke (Nervous system disorders) | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 4 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Parathyroid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 1 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 2 | 0 | 0
Bladder cyst (Renal and urinary disorders) | 0 | 1 | 0
Bladder tamponade (Renal and urinary disorders) | 1 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Pyelectasia (Renal and urinary disorders) | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 1 | 1
Fatigue (General disorders) | 1 | 1 | 0
Catheter related complication (General disorders) | 0 | 0 | 1
Catheter site haemorrhage (General disorders) | 0 | 0 | 1
Hyperthermia (General disorders) | 0 | 0 | 1
Ischaemic ulcer (General disorders) | 0 | 0 | 1
Multi-organ failure (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Sudden death (General disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pneumothorax (General disorders) | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 2 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 1 | 1
Retinal detachment (Eye disorders) | 1 | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Cervix disorder (Reproductive system and breast disorders) | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0
Penile necrosis (Reproductive system and breast disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Cognitive deterioration (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 1
Drug dependence (Psychiatric disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Anaemia vitamin b12 deficiency (Blood and lymphatic system disorders) | 0 | 0 | 1
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 | 0 | 1
Adrenal cortical insufficiency (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RO0503821 (1x/2 Weeks) (N=190) | RO0503821 (1x/4 Weeks) (N=190) | Epoetin Reference (N=191)
Procedural hypotension (Injury, poisoning and procedural complications) | 16 | 28 | 19
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 14 | 15 | 5
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 11 | 13 | 6
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 6 | 11 | 9
Procedural hypertension (Injury, poisoning and procedural complications) | 7 | 13 | 4
Nasopharyngitis (Infections and infestations) | 18 | 19 | 18
Upper respiratory tract infection (Infections and infestations) | 12 | 12 | 11
Bronchitis (Infections and infestations) | 6 | 13 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 | 14 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 8 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 13 | 10
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 11 | 5
Diarrhoea (Gastrointestinal disorders) | 18 | 15 | 14
Abdominal pain upper (Gastrointestinal disorders) | 4 | 11 | 5
Headache (Nervous system disorders) | 15 | 19 | 19
Fluid overload (Metabolism and nutrition disorders) | 9 | 13 | 16
Angina pectoris (Cardiac disorders) | 0 | 13 | 2
Hypertension (Vascular disorders) | 27 | 30 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.